CLINICAL TRIAL: NCT00524186
Title: Phase I Study of Sunitinib With FOLFIRI (Irinotecan, 5-Fluorouracil and Leucovorin) for Advanced Gastroesophageal Cancers
Brief Title: Sunitinib, Irinotecan, Fluorouracil, and Leucovorin In Treating Patients With Advanced Stomach Cancer or Gastroesophageal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left institute
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000562762; RPCI-I-69605
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage III gastric cancer; stage IV gastric cancer; adenocarcinoma of the esophagus; stage IV esophageal cancer; recurrent gastric cancer; recurrent esophageal cancer; adenocarcinoma of the stomach
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Fluorouracil; Irinotecan; Leucovorin; Sunitinib; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral Sunitinib (Experimental): Patients receive oral sunitinib malate on day -7 and then once daily on days 2-28 in course 1 and on days 1-28 in all subsequent courses
  Interventions: Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Drug: sunitinib malate; Other: flow cytometry; Other: pharmacological study

INTERVENTIONS:
Drug: fluorouracil — Given IV
Drug: irinotecan hydrochloride — Given IV
Drug: leucovorin calcium — Given IV
Drug: sunitinib malate — Taken Orally
Other: flow cytometry — Correlative Study
Other: pharmacological study — Correlative Study

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as irinotecan, fluorouracil, and leucovorin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving sunitinib together with combination chemotherapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of sunitinib when given together with irinotecan, fluorouracil, and leucovorin in treating patients with advanced stomach cancer or gastroesophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of sunitinib malate when administered with FOLFIRI chemotherapy comprising irinotecan hydrochloride, fluorouracil, and leucovorin calcium in patients with advanced gastroesophageal cancer.

Secondary

* Determine the response rates, overall survival, and progression-free survival of patients treated with this regimen.
* Determine if there is a change in circulating endothelial precursor cell number and VEGF expression as a result of this therapy and if these changes correlate with improved response and survival.
* Document any pharmacokinetic interactions between irinotecan hydrochloride and sunitinib malate.
* Study pharmacokinetics of sunitinib malate on day 14 (steady state) and day 42 (after 6 weeks of continuous dosing).

OUTLINE: Patients receive oral sunitinib malate on day -7 and then once daily on days 2-28 in course 1 and on days 1-28 in all subsequent courses. Patients also receive FOLFIRI chemotherapy comprising irinotecan hydrochloride IV over 90 minutes, fluorouracil IV continuously over 46 hours, and leucovorin calcium IV over 2 hours beginning on days 1 and 15. Treatment repeats every 4 weeks for up to 12 months in the absence of disease progression or unacceptable toxicity.

Blood is collected at baseline and periodically during study for pharmacokinetic and biomarker correlative studies. Samples are analyzed by flow cytometry to assess circulating endothelial cells and VEGF expression.

After completion of study treatment, patients are followed for 4 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically confirmed diagnosis of 1 of the following:

  * Locally advanced or unresectable gastric cancer
  * Metastatic gastric adenocarcinoma
  * Metastatic gastroesophageal junction (GEJ) adenocarcinoma

    * Esophageal adenocarcinomas with involvement of GEJ allowed

Exclusion criteria:

* Symptomatic, uncontrolled CNS metastases

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-1
* Life expectancy > 12 weeks
* WBC ≥ 3,000/μL
* Platelet count ≥ 100,000/μL
* Creatinine ≤ 1.5 mg/dL
* Bilirubin ≤ 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Exclusion criteria:

* Uncontrolled infection
* Uncontrolled serious medical disease
* Uncontrolled hypertension
* Coagulopathy or bleeding disorder
* History of allergic reactions attributed to compounds of similar chemical or biological composition to sunitinib malate or other agents used in study

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* No prior chemotherapy for metastatic disease
* Concurrent therapeutic anticoagulation allowed

Exclusion criteria:

* Other concurrent investigational therapy
* Concurrent combination antiretroviral therapy in HIV-positive patients
* Major surgery or radiotherapy within the past 3 weeks

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-05; Primary Completion 2013-08 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of sunitinib malate when administered with FOLFIRI chemotherapy (i.e., irinotecan hydrochloride, fluorouracil, and leucovorin calcium) | 30 days after treatment

SECONDARY OUTCOMES:
Toxicity | 28 days
Response rate as assessed by RECIST criteria | Every 3 months up to 5 years
Progression-free survival | Every 3 months up to 5 years
Overall survival | up to 5 years
Circulating endothelial precursor cell (CEC) number | At baseline
VEGF expression | At Baseline
Correlation of pre- and post-therapy changes in CEC number and VEGF expression with response rate and survival | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Boland, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Derived] Mukherjee S, Fountzilas C, Boland PM, Gosain R, Attwood K, Tan W, Khushalani N, Iyer R. Phase I Study of Irinotecan/5-Fluorouracil/Leucovorin (FOLFIRI) with Sunitinib for Advanced Gastric or Gastroesophageal Junction Adenocarcinoma. Target Oncol. 2020 Feb;15(1):85-92. doi: 10.1007/s11523-019-00692-y. PMID 31802410